CLINICAL TRIAL: NCT00678314
Title: Patient Controlled Regional Analgesia Following Carpal Tunnel Release: A Double-Blind Study Using Distal Perineural Catheters
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Dr Kurt Pettersson, Institution for Clinical Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LMV 151:2003/9759
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Anesthetics; Local; ropivacaine; Surgery; Hand; carpel tunnel; Carpal tunnel surgery
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Active Comparator)
  Interventions: Drug: Ropivacaine 0.2%
- Group B (Active Comparator)
  Interventions: Drug: Ropivacaine 0.75%
- Group C (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ropivacaine 0.2% — 10 ml
  Arms: Group A
Drug: Ropivacaine 0.75% — 3 ml
  Arms: Group B
Drug: Normal saline — 10 ml
  Arms: Group C

SUMMARY:
This study was done with the primary aim of assessing the efficacy (as calculated by pain intensity difference) of patient controlled regional analgesia (PCRA) technique against oral analgesics, which has been the standard of care at our hospital. Secondary objectives were to analyze the volume and dose of LA that should be given, patient satisfaction and the long-term outcome for patients treated with the PCRA technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically established carpel tunnel syndrome
* Surgery performed under local anesthesia

Exclusion Criteria:

* Chronic pain requiring analgesics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2004-01; Primary Completion 2006-01 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
This study was done with the primary aim of assessing the efficacy (as calculated by pain intensity difference) of patient controlled regional analgesia (PCRA) technique against oral analgesics, which has been the standard of care at our hospital. | 24 h

SECONDARY OUTCOMES:
Secondary objectives were to analyze the volume and dose of LA that should be given, patient satisfaction and the long-term outcome for patients treated with the PCRA technique. | Up to 1 yr after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Pettersson, MD, PhD, Principal Investigator — Institution for Clinical Medicine
Locations (1):
- Örebro University Hospital, Örebro, Örebro County, Sweden